CLINICAL TRIAL: NCT07194928
Title: Medical Cannabis as an Opiate Alternative
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Franklin Caldera, Professor of Physical Medicine and Rehabilitation, University of Pennsylvania
Other Study IDs: 856134
Record Dates: First submitted 2025-09-11; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain; Opioid Use
Keywords: Chronic pain; Opioid medication; Medical Marijuana
MeSH Terms: conditions — Chronic Pain | interventions — Medical Marijuana

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic opioid pain patients were cost was barrier to trying medical marijuana: Chronic opioid patient who were unable to wean off opioid in the past and unable to try medical marijuana secondary to cost. Patient who are eligible will be certified for their medical marijuana card and will go to dispensary to get their medical marijuana.
  Interventions: Other: We will monitor patient's response to medical marijuana as alternative to opioid for chronic pain.

INTERVENTIONS:
Other: We will monitor patient's response to medical marijuana as alternative to opioid for chronic pain. — We will monitor patient response to medical marijuana as opioid alternative. This will be given to patient who otherwise could not get intervention secondary to cost. We want to show that medical marijuana is a safer alternative to opioids in this population of patients
  Other Names: Medical cannabis

SUMMARY:
Opioid use for pain has increased drastically over last decade with disastrous results that lead to an epidemic of overdoses and deaths in the United States. Philadelphia has been described as "ground zero" in the opiate epidemic of overdoses and deaths in the United States. Some initial clinical experience shows that medical marijuana can potentially assist patients suffering from certain serious medical conditions by alleviating pain and improving quality of life, allowing them to discontinue opiates.

Medical Cannabis is very safe and a viable option for pain relief to improve patients and their family's quality of life. The medical marijuana law in Pennsylvania was passed in 2016 with the hope that this might alleviate the opiate crisis. The opioid death rate in Pennsylvania was 37.9 per 100,000 people. However, medical cannabis is not covered by insurance and is an out of pocket expense. This has been a barrier to some patients trying medical cannabis as an alternative. This can create a disparity in care of chronic pain patients.

Methods:

Recruitment and inclusion/exclusion criteria: Potential participants will be recruited from an outpatient chronic pain clinic. 40 patients who have agreed to attempt wean down on opioid medication and have a diagnosis which qualifies them for medical marijuana will be selected for the study. In these selected patients cost of the treatment was the main barrier for starting medical cannabis. Each participant will undergo a urine drug screen, a pain assessment using the visual analog scale and pain quality will be assessed using the Short Form-36 health related quality and McGill Pain Questionnaire, which measures sensory, affective and evaluative dimensions of pain prior to receiving medical marijuana and then at 6 months.

Each patient will be evaluated by a physician who is certified to evaluate patients for Medical Cannabis. If the patient qualifies for Medical Cannabis the next step is for the patient to register on the state of Pennsylvania medical marijuana website. Medical conditions that qualify patient in the states of Pennsylvania for medical marijuana are Amyotrophic lateral sclerosis, Cancer, Crohn's disease, multiple sclerosis, Neurodegenerative diseases, neuropathies, chronic or intractable pain of neuropathic origin. After the patient registers the physician will also certify them on the website. After the patients are certified they will apply for medical marijuana card. Once the patient receives a medical marijuana card the patient will start an opioid weaning plan. Each patient will have an individualized plan for weaning off their opioids which is their standard care plan. The patient will go to the select medical marijuana dispensary and will be able to choose their medical cannabis product. The Curaleaf medical cannabis dispensary will have a list of patients and participants will be able to choose from the cannabis products. The patient will be followed up monthly for six months by physician and will assess the patient's pain levels and Medical Cannabis doses and opioid doses monthly. The investigators will also note the patient side effects, tolerance and any decrease in symptoms. At six months the physician will recheck a urine drug screen, current pain level and readminister the McGill Pain Questionnaire and Short form-36 health related quality. The Medical Cannabis doses and strains will be noted.

ELIGIBILITY:
Inclusion Criteria:

Patient who are on chronic opioids medication for pain and have failed to wean off in past. These patients also have diagnoses that makes them eligible for medical marijuana and are willing to try it as an alternative to opioids -

Exclusion Criteria: History of Schizophrenia Acute psychiatric disorder Licensed to carry firearm Federal job that excludes them from receiving medical marijuana.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic pain patient on long term opioids who failed to wean off in the past. Patients have no contraindication to medical marijuana and qualify to try as an alternative to opioids.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2024-10-11 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 6 months
  The patient will follow up monthly and have their pain score evaluated monthly morphine, at 1st visit 3rd visit and 6th visit patient will be given McGill Pain evaluation and Short form- 36 questionaire.
Morphine equivalents | 6 months
  The patient will follow up monthly for 6 months and have their morphine equivalent dosing monitored.
McGill Pain evaluation | 1st month, 3rd month and 6th month
  The patient will follow up monthly but McGill Pain questionnaire will be administered at 1st month, 3rd month and 6th month visits.
Short form-36 questionnaire. | 1st month, 3rd month and 6th month
  The patient will follow up monthly but Short Form 36 questionnaire will be administered at 1st month, 3rd month and 6th month visits.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
We only use non identifiable data and do not plan to use any identifiable individual data.

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-10-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT07194928/Prot_ICF_000.pdf